CLINICAL TRIAL: NCT03586765
Title: Assess Prevalence of Urinary Functional Disorders in Women of 40 and More, Visiting a General Practitioner, Occupational Medicine or Health Examination Center in Puy-de-Dôme
Brief Title: Epidemiology of Urinary Functional Disorders in Women of 40 and More
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-395; 2017-A00968-45 (Other: 2017-A00968-45)
Record Dates: First submitted 2018-06-28; First posted 2018-07-16 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Menopause; Overweight; Surgical Antecedent; Gestity
Keywords: incontinence; female; observational study; self filled survey; epidemiology
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental group: Assess prevalence of urinary functional disorders in women of 40 and more, visiting a general practitioner, occupational medicine or health examination center in Puy-de-Dôme. Study conducted for a month using a self-filled survey distributed by secretaries or nurses.
  Interventions: Other: Female urinary incontinence

INTERVENTIONS:
Other: Female urinary incontinence — Assess prevalence of urinary functional disorders in women of 40 and more, visiting a general practitioner, occupational medicine or health examination center in Puy-de-Dôme. Study conducted for a month using a self-filled survey distributed by secretaries or nurses.

SUMMARY:
Assess prevalence of urinary functional disorders in women of 40 and more, visiting a general practitioner, occupational medicine or health examination center in Puy-de-Dôme. Study conducted for a month using a self-filled survey distributed by secretaries or nurses.

DETAILED DESCRIPTION:
The diagnosis of urinary incontinence is clinical. Three types of urinary incontinence are described: urinary stress incontinence, urinary incontinence by overactive bladder or mixed urinary incontinence.

To standardize the medical examination and to precise the urinary incontinence type, the use of a validated questionnaire is recommended (USP), the quality of life's resounding also must be assessing, using questionnaire of quality of life valid in French (ICIQ®, CONTILIFE®…) Several medical cares exist, but patients often don't know it. Unhappily, it is still a taboo subject. In a French medical study, conducted in 1992 by 60 general practitioners, of a total of 2911 female patients, 37% said they had urinary disorders. Among them, 77% said they had symptoms during an effort, 57% had urinary urge incontinence and 35 % had spontaneous leaks. One in five women had three associated disorders.

In a French study conducted in 2005, it appeared that women talked to their general practitioner about urinary disorders only four or five times out of ten, and six times out of ten when they used panty liners.

The results are eloquent, but the data is not recent, and the investigators need some, to propose better cares.

This medical study will be conducted during one month. Two self-filled questionnaires will be distributed by nurses or medical secretary, working at recruited general practitioner's place, to every female patient who will be 40 years old or more, coming for themselves or accompanying somebody else (children for example). Every female patient will have to fill both questionnaires alone, anonymously, and will have to let them in a closed box, in the waiting room.

The two self-filled questionnaires are called USP and CONTILIFE. They are both validated to evaluate symptoms and quality of life.

Additional question about existence of fecal incontinence (and its type), and the reasons why patients didn't talk about it with their general practitioner spontaneously (shame, absence of information about cares, fatality…).

Prior visit of each recruited service by Julie de la Roque, to explain the goals of the study, to general practitioners, nurses and medical secretaries.

ELIGIBILITY:
Inclusion Criteria:

* female
* 40 and more
* speaking French

Exclusion Criteria:

* men
* female of less than 40
* not speaking French
* refusal
* inability to answer questions

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: women of 40 and more
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
current urinary functional disorders prevalence in women of 40 and more | between november 13th, 2017 and december 15th, 2017
  A difference will be made between urinary stress incontinence and overactive bladder. Each disorder is characterized by a score (not available for patients). The doctor will calculate the score for each one ( from 0 to 9 for urinary stress incontinence, and from 0 to 21 for urinary incontinence by overactive bladder ). A disorder will be considered positive if it is greater than or equal to 1.

SECONDARY OUTCOMES:
Relationship between age and occurrence of functional urinary disorders for same aged groups | between november 13th, 2017 and december 15th, 2017
  question on the self-filled
Relationship between menopause and occurrence of functional urinary disorders for same aged groups | between november 13th, 2017 and december 15th, 2017
  question on the self-filled
Relationship between childbirth way (caesarean or natural way) and occurrence of functional urinary disorders | between november 13th, 2017 and december 15th, 2017
  question on the self-filled
Relationship between carrying of loads within the framework of the occupation and occurrence of functional urinary disorders | between november 13th, 2017 and december 15th, 2017
  question on the self-filled
Relationship between dwelling place and occurrence of functional urinary disorders | between november 13th, 2017 and december 15th, 2017
  question on the self-filled

CONTACTS AND LOCATIONS:
Overall Officials: Julie DE LA ROQUE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont-Ferrand, Clermont-Ferrand, France